CLINICAL TRIAL: NCT07202403
Title: Iterative Design Trial to Assess Dietary Supplements and Other Aging-targeted Therapies
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Atria Research and Global Health Institute (ARGHI) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: #25-02-400-2231
Record Dates: First submitted 2025-09-02; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Aging; Longevity
Keywords: spermidine; aging; longevity; healthspan
MeSH Terms: interventions — Spermidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spermidine (Experimental): Participants will receive capsules for three consecutive 28-day courses with escalating doses of 40mg, 120mg, and 400mg.
  Interventions: Dietary Supplement: Spermidine

INTERVENTIONS:
Dietary Supplement: Spermidine — Spermidine is a polyamine that forms naturally in plants, animals, and microorganisms as a byproduct of protein breakdown. While it's found in various foods, the highest concentrations are in wheat germ, soy, and fermented foods like cheese and miso (Madeo et al. 2018). Spermidine is known for its role in promoting autophagy, a cellular process that helps to clear damaged cells and improve overall cellular function (Eisenberg et al. 2009; Gabandé-Rodríguez, Gómez de Las Heras, and Mittelbrunn 2019). As a result, spermidine has recently attracted significant scientific interest for its potential to enhance lifespan and overall health in laboratory studies.

SUMMARY:
This is a multi-cohort, open-label, adaptive trial designed to evaluate the safety, tolerability, and biological effects of dietary supplements and other aging-targeted therapies.

Cohort 1 is a single-arm, open-label, intrapatient dose-escalation study evaluating the effects of escalating doses of spermidine in 10 participants. Patients will have baseline blood drawn and subsequently start daily administration of spermidine. They will receive capsules for three consecutive 28-day courses with escalating doses of 40mg, 120mg, and 400mg.

Subsequent cohorts will evaluate additional agents.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 75
* Patients without known significant organ dysfunction, based on standard blood tests within the last year

Exclusion Criteria:

* Patients taking any immunomodulatory medications that the investigator or treating physician believe may alter the immune response to the study agent (e.g. biologic antibodies, immunosuppressants)
* Patients actively receiving any therapy that, in the determination of the investigator, may impact the effect of the study agent.
* Patients who, in the opinion of the treating investigator, will not be able to follow treatment and defined follow-up
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2030-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Baseline to Day 112
  Assessment of toxicity of therapeutic intervention. Toxicity will be assessed through adverse event monitoring conducted at clinic visits or by phone, with adverse events evaluated and graded using CTCAE v5.0.

SECONDARY OUTCOMES:
Change in systemic immune milieu | Baseline and approximately every 28 days through Day 112 (final study visit).
  Change in circulating immune biomarkers from baseline and across dose levels, including cytokines and chemokines and immune cell subsets.
Change in systemic metabolic milieu | Baseline and approximately every 28 days through Day 112 (final study visit).
  Metabolomics profiling to quantify circulating plasma metabolites and assess dynamic changes at each dose level.

CONTACTS AND LOCATIONS:
Locations (1):
- Atria Research and Global Health Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
To safeguard participant privacy, only fully de-identified data may be shared with qualified researchers under appropriate data use agreements and in compliance with all applicable privacy regulations.